CLINICAL TRIAL: NCT00334984
Title: Prevention of Mucositis in Children With AES-14 (IND#36978), a Glutamine Based Oral Care Regimen, for Patients Diagnosed With Solid Tumors: A Randomized Placebo-Controlled Clinical Study
Brief Title: Glutamine in Preventing Oral Mucositis in Patients Receiving Chemotherapy for Sarcoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to inability to reach an acceptable agreement with industry sponsor
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: ANUR0532; COG-ANUR0532; CDR0000469005
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Childhood Malignant Fibrous Histiocytoma of Bone; Sarcoma
Keywords: childhood fibrosarcoma; childhood neurofibrosarcoma; childhood synovial sarcoma; chondrosarcoma; localized osteosarcoma; metastatic osteosarcoma; metastatic childhood soft tissue sarcoma; nonmetastatic childhood soft tissue sarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; localized Ewing sarcoma/peripheral primitive neuroectodermal tumor; previously treated childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; childhood alveolar soft-part sarcoma; childhood angiosarcoma; childhood epithelioid sarcoma; childhood leiomyosarcoma; childhood liposarcoma; localized childhood malignant fibrous histiocytoma of bone; metastatic childhood malignant fibrous histiocytoma of bone; childhood malignant mesenchymoma; dermatofibrosarcoma protuberans; childhood desmoplastic small round cell tumor
MeSH Terms: conditions — Sarcoma; Fibrosarcoma; Chondrosarcoma; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Hemangiosarcoma; Liposarcoma; Malignant mesenchymal tumor; Dermatofibrosarcoma; Desmoplastic Small Round Cell Tumor | interventions — Glutamine

INTERVENTIONS:
Drug: glutamine
Procedure: chemoprotection
Procedure: management of therapy complications
Procedure: therapeutic nutritional supplementation

SUMMARY:
RATIONALE: Glutamine may help prevent mucositis, or mouth sores, in patients receiving chemotherapy for sarcoma. It is not yet known whether glutamine is more effective than a placebo in preventing mucositis in patients receiving chemotherapy for sarcoma.

PURPOSE: This randomized clinical trial is studying glutamine to see how well it works compared to a placebo in preventing oral mucositis in patients receiving chemotherapy for sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of a new preparation of glutamine (AES-14) vs placebo in reducing the incidence of grade 3 or 4 chemotherapy-induced oral mucositis during the first course of chemotherapy in patients with sarcomas.

Secondary

* Compare the rates of mucositis-related chemotherapy dose reductions for the subsequent course of anthracycline-based chemotherapy in patients treated with AES-14 vs placebo.
* Compare the rates of mucositis-related delays of chemotherapy administration for the next chemotherapy course in patients treated with AES-14 vs placebo.
* Compare the rates of systemic and oral infections during the first course of chemotherapy in patients treated with AES-14 vs placebo.
* Compare the number of days of narcotic use for mucositis-related pain during the first course of chemotherapy in patients treated with AES-14 vs placebo.
* Determine the inter-rater reliability between caregivers and nurses in the use of the modified Walsh scale.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to age (5-10 years vs 11-18 years vs 19-30 years) and diagnosis (Ewing's sarcoma vs osteogenic sarcoma vs rhabdomyosarcoma vs other sarcomas). Patients are randomized to 1 of 2 treatment arms.

* Arm I (glutamine [AES-14]): Patients rinse with oral AES-14 for at least 30 seconds and then swallow (swish and swallow) three times daily beginning on the day of or within 1 day before starting their first course of chemotherapy. Patients also undergo a standard oral care regimen comprising brushing their teeth at least twice daily, 30 minutes or more after taking AES-14, and rinsing with water at least twice daily. Treatment continues until blood counts recover and patient's total modified Walsh score ≤ 2 (mucositis score).
* Arm II (placebo): Patients swish and swallow oral placebo and undergo a standard oral care regimen as in arm I.

Caregivers assess the patient's mouth daily while the patient is receiving the study drug. Caregivers keep a daily diary rating the patient's oral mucosal areas and degree of pain, describing the patient's oral intake, and documenting that the study drug was used and standardized oral care was performed.

PROJECTED ACCRUAL: A total of 180 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with any of the following:

  * Ewing's sarcoma
  * Osteogenic sarcoma
  * Rhabdomyosarcoma
  * Other sarcomas (i.e., fibrosarcoma or synovial sarcoma)
* Scheduled to receive first course of chemotherapy that includes ≥ 75 mg/m² of anthracyclines
* Total modified Walsh score ≤ 2 (mucositis score)

PATIENT CHARACTERISTICS:

* Must have a caregiver (parent, other relative, or friend) available to perform daily mucositis assessments
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 5 times ULN
* Albumin ≥ 2 g/dL
* No history of hypersensitivity to any known component of AES-14

PRIOR CONCURRENT THERAPY:

* No prior glutamine (AES-14)
* No prior or concurrent head and/or neck radiation therapy
* No concurrent supplementation with another glutamine product
* No other concurrent agents for mucositis prophylaxis

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Donna L. Betcher, RN, MSN, Study Chair — Mayo Clinic